CLINICAL TRIAL: NCT01131871
Title: Enhanced Behavioral Intervention to Improve Long-Term Weight Loss in Young Adults
Brief Title: Innovative Approaches to Diet, Exercise and Activity
Acronym: IDEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, John M. Jakicic, PhD, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01HL096770 (NIH)
Record Dates: First submitted 2010-05-24; First posted 2010-05-27 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Body Weight
Keywords: obesity; overweight
MeSH Terms: conditions — Body Weight; Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Behavioral Weight Loss Intervention (Active Comparator)
  Interventions: Behavioral: Standard Behavioral Weight Loss Intervention
- Enhanced Weight Loss Intervention (Experimental)
  Interventions: Behavioral: Enhanced Weight Loss Intervention

INTERVENTIONS:
Behavioral: Standard Behavioral Weight Loss Intervention — Subjects in this group will receive our standard behavioral weight control program that is delivered in an in-person group-based format. At month 7 subjects will also be given access to a study website to monitor eating and activity behaviors, and to have electronic access to standardized intervention materials. At month 7 subjects will also receive targeted study-related text messages that otherwise would have been provided in paper format.
  Arms: Standard Behavioral Weight Loss Intervention
Behavioral: Enhanced Weight Loss Intervention — Subjects in this group will participate in a weight loss intervention that includes technology enhancements. These enhancements will include the addition of intervention specific targeted and tailored text messaging and the BodyMedia Fit System® beginning at Month 7. At month 7 subjects in EWLI will also receive the same targeted study-related text messages provided to SBWP that otherwise would have been provided in paper format.
  Arms: Enhanced Weight Loss Intervention

SUMMARY:
The prevalence of obesity in young adults has been increasing, and excessive body weight have been linked to numerous chronic conditions including cardiovascular disease, diabetes, many forms of cancer, and numerous musculoskeletal problems. This study will focus of the development and evaluation of interventions that may be appropriate for young adults (age 18-35 years) to improve weight loss outcomes following a 24 month intervention. The primary aim of this study is to examine whether an enhanced weight loss intervention (EWLI) that includes technology components results in improved weight loss in young adults (18-35 years of age) compared to a standard behavioral weight loss intervention (SBWP) over a period of 24 months. Eligible participants will also be assessed for body composition, body fat distribution, fitness, physical activity, dietary intake, and behavioral/psychosocial measures that may be predictive of behavior change. Assessments will occur at 0, 6, 12, 18, and 24 months. Subjects will participate in a 24 month behavioral weight loss program that includes a reduction in energy intake and moderate-to-vigorous intensity exercise (progressively increasing from 100 to 300 minutes per week). The technologies added to EWLI are text messaging, a wearable device that provides feedback on physical activity, and access to a website to monitor dietary behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age
* Intending to be available for a 24 month intervention
* An active cellular telephone that is capable of receiving text messaging
* A computer and internet connectivity that can be used for the BodyMedia Fit system
* Body mass index (BMI) between 25.0-39.9 kg/m2
* The ability to provide medical clearance to participate in this study from their primary care physician
* The ability to complete the baseline graded exercise test, and clearance from the study physician to participate in this study after reviewing the results from this study

Exclusion Criteria:

* Unable to provide informed consent
* Household member on study staff
* Past or planned (within the next 24 months) weight loss surgery (e.g. gastric bypass, lap band, or liposuction); current participation in a commercial weight loss program (e.g. Weight Watcher's, Jenny Craig); current or planned enrollment in another diet/PA/weight loss intervention study
* Report regular use of systemic steroids, prescription weight loss drugs. "Regular use" is defined as "taking this medication most days of the week for the previous month"
* Current treatment for eating disorder
* Cardiovascular event (heart attack, stroke, episode of heart failure, or revascularization procedure) within the last 6 months
* Current treatment for malignancy (other than non-melanoma skin cancer)
* Currently pregnant or gave birth within the last 6 months, currently lactating or breastfeeding within the last 3 months, actively planning pregnancy within the next 24 months
* Investigator discretion
* Currently taking medication that would affect heart rate or blood pressure responses to exercise (e.g., beta blockers)
* Report losing >5% of current body weight in the previous 6 months
* Currently treated for psychological issues, or taking psychotropic medications within the previous 6 months
* Report taking medication that could affect metabolism or change body weight
* Current treatment for diabetes mellitus

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 471 (Actual)
Dates: Start 2010-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
weight change | Change from baseline to 24 months
  Body weight will be assessed on a digital scale to assess change in body weight over the 24 month intervention period.

SECONDARY OUTCOMES:
body composition | 0, 6, 12, 18 24 months
  Body composition will be assessed using DXA. This will provide a measure of lean body mass, fat mass, bone mineral content, and percent body fat.
cardiorespiratory fitness | 0, 6, 12, 18, 24 months
  A graded exercise test on a treadmill along with indirect calorimetry will be used to measure cardiorespiratory fitness. This will provide a measure of oxygen consumption and metabolic equivalents of work at the time of test termination.
physical activity energy expenditure | 0, 6, 12, 18, 24 months
  A questionnaire and a portable device worn on the upper arm will be used to measure and quantify energy expenditure from physical activity.
dietary intake | 0, 6, 12, 18, 24 months
  A questionnaire will be used to assess self-reported food intake. This will be used to estimate calories, dietary fat, protein, and carbohydrates consumed.
psychosocial and behavioral measures | 0, 6, 12, 18, 24 months
  Questionnaires will be used to assess self-efficacy for weight loss and physical activity, barriers to physical activity and weight loss, expected outcomes resulting from physical activity and weight loss, perceived body image, depressive symptomotology, sleep patterns, weight history, dietary disinhibition and restraint, and behaviors typically related to weight loss (e.g., self-weighing, meal planning, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: John M Jakicic, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jakicic JM, Davis KK, Rogers RJ, King WC, Marcus MD, Helsel D, Rickman AD, Wahed AS, Belle SH. Effect of Wearable Technology Combined With a Lifestyle Intervention on Long-term Weight Loss: The IDEA Randomized Clinical Trial. JAMA. 2016 Sep 20;316(11):1161-1171. doi: 10.1001/jama.2016.12858. PMID 27654602
- [Derived] Jakicic JM, King WC, Marcus MD, Davis KK, Helsel D, Rickman AD, Gibbs BB, Rogers RJ, Wahed A, Belle SH. Short-term weight loss with diet and physical activity in young adults: The IDEA study. Obesity (Silver Spring). 2015 Dec;23(12):2385-97. doi: 10.1002/oby.21241. Epub 2015 Nov 5. PMID 26538477
- [Derived] Jakicic JM, King WC, Gibbs BB, Rogers RJ, Rickman AD, Davis KK, Wahed A, Belle SH. Objective Versus Self-Reported Physical Activity in Overweight and Obese Young Adults. J Phys Act Health. 2015 Oct;12(10):1394-400. doi: 10.1123/jpah.2014-0277. Epub 2015 Jan 19. PMID 25599334